CLINICAL TRIAL: NCT04216940
Title: Assessment of Pain Intensity After Instrumentation by MPRo and Hyflex Rotatry Files in Molars With Irreversible Pulpitis
Brief Title: Pain Intensity After Root Canal Instrumentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Maram Obeid, Ass. Prof., Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: pain intensity
Record Dates: First submitted 2019-12-24; First posted 2020-01-03 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2020-01

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- M-pro (Experimental)
  Interventions: Device: mechanical preparation of root canal system
- Hyflex (Experimental)
  Interventions: Device: mechanical preparation of root canal system

INTERVENTIONS:
Device: mechanical preparation of root canal system — Assess the pain intensity in a two-visit treatment of molars with irreversible pulpitis after instrumentation with two different rotary Nickle Titanium systems

SUMMARY:
Assess the pain intensity in a two visit treatment of molars with irreversible pulpitis after instrumentation with two rotary systems Mpro and Hyflex files.

ELIGIBILITY:
Inclusion Criteria:

* mandibular molars with acute pulpitis

Exclusion Criteria:

* badly decayed non-restorable molars
* medically compromised patients

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2019-02-10 (Actual); Primary Completion 2019-08-28 (Actual); Study Completion 2019-08-28 (Actual)

PRIMARY OUTCOMES:
Pain felt after mechanical instrumentation in the first visit | up to 72 hours
  using Numeric Rating Scale (NRS) the participant will be asked to verbally rate their pain on a scale from 0 to 10, with 0 equal to no pain and 10 equal to worst possible pain

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt